CLINICAL TRIAL: NCT03918356
Title: Application of Electrical Impedance Myography (EIM) to Establish Muscle Impedance Parameters as a Potential Biomarker of Idiopathic Inflammatory Myopathies (IIMs)
Brief Title: Application of Electrical Impedance Myography (EIM) as a Potential Biomarker of Idiopathic Inflammatory Myopathies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 2000024786
Record Dates: First submitted 2019-04-12; First posted 2019-04-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inclusion Body Myositis patients (Experimental): Subjects with clinically or clinico-pathologically defined IBM will be included in this study. Patients with consistent clinical and laboratory features including ages 18 to 80 years, duration of symptoms> 12 months, serum creatine kinases (CK) no greater than 15 times upper limit of normal, prominent weakness of quadriceps and/or finger flexor weakness>shoulder abduction weakness along with some characteristic histopathological findings of endomysial inflammatory infiltrate, rimmed vacuoles and protein accumulation or 15-18 nm filaments will be considered as clinically or clinicopathologically defined IBM as proposed by the European Neuromuscular Center (ENMC IBM working group, 2013).
  Interventions: Device: electrical impedance myography
- Idiopathic Inflammatory Myopathies patients (Experimental): Subjects with more than 2 of the following criteria, symmetric proximal weakness, elevated CK, electromyography (EMG) suggesting myositis, muscles biopsy showing inflammatory changes, and typical skin rashes of dermatomyositis (DM) will be recruited as dermatomyositis and polymyositis (DM/PM) based on Bohan and Peter criteria.
  Interventions: Device: electrical impedance myography
- control (Placebo Comparator): Healthy controls without any known neuromuscular disorders and no family history of Amyotrophic lateral sclerosis (ALS) will be recruited for the study.
  Interventions: Other: healthy control group

INTERVENTIONS:
Device: electrical impedance myography — Electrical impedance myography (EIM) is a new electrodiagnostic method of quantitative muscle evaluation. It utilizes concepts of bio impedance, the ability of biological tissue to impede externally applied electrical current.
  Arms: Idiopathic Inflammatory Myopathies patients; Inclusion Body Myositis patients
Other: healthy control group — healthy control
  Arms: control

SUMMARY:
1. To assess changes in impedance parameters in Idiopathic Inflammatory Myopathies (IIMs).
2. To assess whether EIM parameters are reflective of disease severity, based on clinical outcome measures of IIMs.

DETAILED DESCRIPTION:
1. To assess changes in impedance parameters in Idiopathic Inflammatory Myopathies (IIMs) There are structural and compositional changes in muscles, such as edema, adipose infiltration, and/or atrophy, in IIMs. Electrical impedance myography (EIM) is sensitive to such changes. EIM parameters will be different when compared to healthy controls in IIMs.
2. To assess whether EIM parameters are reflective of disease severity, based on clinical outcome measures of IIMs.

Clinical outcome measures reflect on disease severity which is an indirect measure of muscle involvement in IIMs. If EIM parameters correlate with clinical outcome measure, it would indirectly prove that EIM can reflect disease severity in IIMs

ELIGIBILITY:
Inclusion Criteria:

* duration of weakness >12 months.
* ages 18 to 80 years old.
* serum CK level no greater than 15 times the upper limit of normal.
* quadriceps weakness >hip flexor weakness and/or finger flexor weakness >shoulder abduction weakness.
* one or more of the following pathological findings:
* endomysial inflammatory infiltrate.
* rimmed vacuoles.
* protein accumulation or 15-18 mm filaments.

DM/PM inclusion criteria:

* ages 18 to 80
* Symmetric proximal weakness
* Elevated CK
* EMG suggestive of myopathy with evidence of muscle membrane irritation
* Muscle biopsy suggestive of inflammatory myositis (degeneration, regeneration, necrosis, and interstitial mononuclear infiltrates)
* Typical skin rashes of DM (Heliotrope rash or Gottron sign)

Key inclusion criteria for the control group:

* no active neuromuscular disorders or known history of neuromuscular disorders.
* no sign or symptoms of muscle weakness.
* no family history of muscular dystrophies or ALS.
* ages 18 to 80

Exclusion Criteria:

* Patients with decompensated congestive heart failure
* Patients with chronic kidney disease on hemodialysis
* Patients with active cancer on chemotherapy or radiotherapy
* Patients with severe disease who are already wheel chair bound

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Manual Muscle Testing Score | 2 years
  This scale reflects on muscle strength. It is based on Medical Research Council scale for muscle power, where muscle strength can have a score of 0-5 (0 means no strength and 5 means full strength).Several muscles are examined in Manual Muscle Testing (MMT) and the total strength is reported as the sum of the Medical Research Council (MRC) muscles scale score of each muscles. Total MMT score for this study can range from 0-160, where 0 means no strength in any muscles and 160 means full strength in all the muscles examined.
IBM-Functional rating scale (IBM-FRS) | 2 years
  This scale measure the limitations in daily life from IBM. It ask 10 questions regarding the activities of daily life and each question is scored between 0-4 (Where 4 means no difficulty and 0 means maximum difficulty). Total score can vary from 0-40, and 40 means no limitations in daily life from IBM.
Grip test | 2 years
  A change in grip strength using a Jamar hand dynamometer to assess the grip strength in every participant. Best of three attempts will be used.
Get up and go test | 2 years
  Time will be measured for a participant to stand up from a chair (using arms if necessary), walk 3 meters, turn around, return to the chair, and sit down. The better of two trials will be used.
Six minute walk | 2 years
  Distance walked in 6 minutes will be measured. This has been used as a primary and secondary outcome measures in several clinical trials in various neuromuscular disorders.
Quality of Health and Well Being | 2 years
  Short Form-36 (SF-36) is a measure of the global quality of health and well-being. The SF-36 is an eight-scaled score, which are the weighted sums of the questions in their corresponding section. Each scale can be transformed into a 0-100 scale. Lower score means more disability.
  SF-36 will be scored utilizing a standardized scoring manual. We will obtain a physical component summary scale and a mental component summary scale.
Myositis Intention to Treat Activities Index (MITAX) | 2 years
  MITAX is a scale assessing the extra-muscular disease severity of myositis. It contains 24 questions covering 7 extra muscular organ systems. Each question is scored between 0-4, where 0 = not present, 1= improving, 2= same, 3= worse, and 4= new. This score is then converted to a final score ranging from A-E for each system based on a predefined scoring schema. Total MITAX score can range between 0 to 54.
Physician Global Assessment Score | 2 years
  This is recorded on a 10-cm visual analog scale (VAS) by the physician at the time of evaluation. The score should reflect on the individual's appearance, medical history, physical examination, laboratory testing, and prescribed medical therapy. In this scale 0 means no evidence of disease related damage and 10 means extremely severe damage.

CONTACTS AND LOCATIONS:
Overall Officials: Bhaskar Roy, MD, Principal Investigator — Yale University
Locations (1):
- Bhaskar Roy, New Haven, Connecticut, United States